CLINICAL TRIAL: NCT05380648
Title: Predicting Outcome of Total Knee Replacement Surgery in Patients With Knee Osteoarthritis: a Prospective Study on the Role of Altered Central Pain Processing and Structural, Functional, Metabolic, Inflammatory and Psychological Factors
Brief Title: Predicting Outcome of Total Knee Replacement Surgery in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Sophie Vervullens, Doctoral student Sophie Vervullens, Universiteit Antwerpen
Other Study IDs: 13/47/472
Record Dates: First submitted 2021-04-29; First posted 2022-05-19 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty surgery will be performed by different orthopedist.

SUMMARY:
Osteoarthritis (OA) is the main cause of pain and disability in elderly. For knee OA, a total knee replacement (TKR) is an effective surgical treatment, and the majority of patients report substantial pain relief and functional improvement following surgery. However, 20-40% of patients undergoing TKR are dissatisfied with postsurgical outcome. Even after revision, some patients keep complaining of persisting pain.

In this study, the investigators will examine putative prognostic factors on the basis of the biopsychosocial model. Besides several psychological factors (measured with questionnaires), the investigators will assess structural impairments (such as radiographic severity of OA), functional impairments (muscle weakness and proprioceptive deficits), anesthetic procedures, immediate postoperative pain management, metabolic factors (body composition and hemoglobin A1c), inflammatory factors (C-Reactive Protein) and the investigators also will examine the role of altered central pain processing (CPP) (primary and secondary mechanical hyperalgesia, mechanical temporal summation, thermal primary and secondary hyperalgesia, endogenous pain modulation).

With a longitudinal study design, this study will explore which factors are predictive of poor outcome in knee OA patients after TKR. Moreover, the interrelationship between CPP, structural, functional, metabolic, inflammatory and psychological factors, and the clinical expression of knee OA (pain, symptoms, physical performance and quality of life) will be investigated.

Further research on the role of the aforementioned putative prognostic factors on postsurgical outcome could contribute to better management of these patients, since these factors may be particularly important for patient-tailored treatment.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA patients >40 years awaiting TKR surgery. Both men and women of all ethnical backgrounds are included.

Exclusion Criteria:

* Patients with diagnosis of neurological/ systemic diseases, possibly impacting pain
* Patients who are not capable of understanding and speaking Dutch
* Revision surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee OA patients awaiting primary TKR surgery will be recruited at the University Hospital of Antwerp (BE), AZ Monica (BE), the academic hospital of Maastricht (NL) and St Jans Gasthuis Weert (NL). In each hospital, at least one orthopaedic surgeon already agreed to participate in this study and to recruit patients.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline pain intensity at 3 months postoperative
  The subscale 'Pain' of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome measure. Minimum score is 0, maximum score is 36. Scores are always transformed to a 0-100 scale. The higher the score, the higher the pain intensity.
Pain intensity | Change from baseline pain intensity at 1 year postoperative
  The subscale 'Pain' of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome measure. Minimum score is 0, maximum score is 36. Scores are always transformed to a 0-100 scale. The higher the score, the higher the pain intensity.
Pain intensity | Change from 3 months postoperative at 1 year postoperative
  The subscale 'Pain' of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome measure. Minimum score is 0, maximum score is 36. Scores are always transformed to a 0-100 scale. The higher the score, the higher the pain intensity.
Pain intensity | Baseline (preoperative)
  The subscale 'Pain' of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome measure. Minimum score is 0, maximum score is 36. Scores are always transformed to a 0-100 scale. The higher the score, the higher the pain intensity.
Pain intensity | 3 months postoperative
  The subscale 'Pain' of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome measure. Minimum score is 0, maximum score is 36. Scores are always transformed to a 0-100 scale. The higher the score, the higher the pain intensity.
Pain intensity | 1 year postoperative
  The subscale 'Pain' of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome measure. Minimum score is 0, maximum score is 36. Scores are always transformed to a 0-100 scale. The higher the score, the higher the pain intensity.

SECONDARY OUTCOMES:
Central pain processing: mechanical local and widespread hyperalgesia allodynia | Change from baseline (preoperative) to 3 months postoperative
  Measured with quantitative sensory testing (QST): mechanical pain pressure threshold measured with digital algometer at the medial knee joint line, lateral knee joint line and m. Tibialis anterior of affected leg, m. extensor carpi radialis of non-dominant arm and forehead.
Central pain processing: mechanical local and widespread hyperalgesia allodynia | Change from baseline (preoperative) to 1 year postoperative
  Measured with quantitative sensory testing (QST): mechanical pain pressure threshold measured with digital algometer at the medial knee joint line, lateral knee joint line and m. Tibialis anterior of affected leg, m. extensor carpi radialis of non-dominant arm and forehead.
Central pain processing: mechanical local and widespread hyperalgesia allodynia | Change from 3 months postoperative to 1 year postoperative
  Measured with quantitative sensory testing (QST): mechanical pain pressure threshold measured with digital algometer at the medial knee joint line, lateral knee joint line and m. Tibialis anterior of affected leg, m. extensor carpi radialis of non-dominant arm and forehead.
Central pain processing: mechanical local and widespread hyperalgesia allodynia | Baseline (preoperative)
  Measured with quantitative sensory testing (QST): mechanical pain pressure threshold measured with digital algometer at the medial knee joint line, lateral knee joint line and m. Tibialis anterior of affected leg, m. extensor carpi radialis of non-dominant arm and forehead.
Central pain processing: mechanical local and widespread hyperalgesia allodynia | 3 months postoperative
  Measured with quantitative sensory testing (QST): mechanical pain pressure threshold measured with digital algometer at the medial knee joint line, lateral knee joint line and m. Tibialis anterior of affected leg, m. extensor carpi radialis of non-dominant arm and forehead.
Central pain processing: mechanical local and widespread hyperalgesia allodynia | 1 year postoperative
  Measured with quantitative sensory testing (QST): mechanical pain pressure threshold measured with digital algometer at the medial knee joint line, lateral knee joint line and m. Tibialis anterior of affected leg, m. extensor carpi radialis of non-dominant arm and forehead.
Central pain processing: bottom-up sensitization | Change from baseline (preoperative) to 3 months postoperative
  Measured with quantitative sensory testing (QST): temporal summation measured with a 60g Von Frey monofilament at the medial knee and lateral knee of affected leg, dorsal wrist of affected side
Central pain processing: bottom-up sensitization | Change from baseline (preoperative) to 1 year postoperative
  Measured with quantitative sensory testing (QST): temporal summation measured with a 60g Von Frey monofilament at the medial knee and lateral knee of affected leg, dorsal wrist of affected side
Central pain processing: bottom-up sensitization | Change from 3 months postoperative to 1 year postoperative
  Measured with quantitative sensory testing (QST): temporal summation measured with a 60g Von Frey monofilament at the medial knee and lateral knee of affected leg, dorsal wrist of affected side
Central pain processing: bottom-up sensitization | Baseline (preoperative)
  Measured with quantitative sensory testing (QST): temporal summation measured with a 60g Von Frey monofilament at the medial knee and lateral knee of affected leg, dorsal wrist of affected side
Central pain processing: bottom-up sensitization | 3 months postoperative
  Measured with quantitative sensory testing (QST): temporal summation measured with a 60g Von Frey monofilament at the medial knee and lateral knee of affected leg, dorsal wrist of affected side
Central pain processing: bottom-up sensitization | 1 year postoperative
  Measured with quantitative sensory testing (QST): temporal summation measured with a 60g Von Frey monofilament at the medial knee and lateral knee of affected leg, dorsal wrist of affected side
Central pain processing: Thermal hyperalgesia | Change from baseline (preoperative) to 3 months postoperative
  Measured with quantitative sensory testing (QST): thermal pain sensitivity measured with thermal rollers (Rolltemp II somedic senselab) at the medial knee and lateral knee of affected leg and m. extensor carpi radialis of non-dominant arm.
Central pain processing: Thermal hyperalgesia | Change from baseline (preoperative) to 1 year postoperative
  Measured with quantitative sensory testing (QST): thermal pain sensitivity measured with thermal rollers (Rolltemp II somedic senselab) at the medial knee and lateral knee of affected leg and m. extensor carpi radialis of non-dominant arm.
Central pain processing: Thermal hyperalgesia | Change from 3 months postoperative to 1 year postoperative
  Measured with quantitative sensory testing (QST): thermal pain sensitivity measured with thermal rollers (Rolltemp II somedic senselab) at the medial knee and lateral knee of affected leg and m. extensor carpi radialis of non-dominant arm.
Central pain processing: Thermal hyperalgesia | Baseline (preoperative)
  Measured with quantitative sensory testing (QST): thermal pain sensitivity measured with thermal rollers (Rolltemp II somedic senselab) at the medial knee and lateral knee of affected leg and m. extensor carpi radialis of non-dominant arm.
Central pain processing: Thermal hyperalgesia | 3 months postoperative
  Measured with quantitative sensory testing (QST): thermal pain sensitivity measured with thermal rollers (Rolltemp II somedic senselab) at the medial knee and lateral knee of affected leg and m. extensor carpi radialis of non-dominant arm.
Central pain processing: Thermal hyperalgesia | 1 year postoperative
  Measured with quantitative sensory testing (QST): thermal pain sensitivity measured with thermal rollers (Rolltemp II somedic senselab) at the medial knee and lateral knee of affected leg and m. extensor carpi radialis of non-dominant arm.
Central pain processing: dysfunctional endogenous pain analgesia | Change from baseline (preoperative) to 3 months postoperative
  Measured with quantitative sensory testing (QST): conditioned pain modulation measured Medoc at both wrists
Central pain processing: dysfunctional endogenous pain analgesia | Change from baseline (preoperative) to 1 year postoperative
  Measured with quantitative sensory testing (QST): conditioned pain modulation measured Medoc at both wrists
Central pain processing: dysfunctional endogenous pain analgesia | Change from 3 months postoperative to 1 year postoperative
  Measured with quantitative sensory testing (QST): conditioned pain modulation measured Medoc at both wrists
Central pain processing: dysfunctional endogenous pain analgesia | Baseline (preoperative)
  Measured with quantitative sensory testing (QST): conditioned pain modulation measured Medoc at both wrists
Central pain processing: dysfunctional endogenous pain analgesia | 3 months postoperative
  Measured with quantitative sensory testing (QST): conditioned pain modulation measured Medoc at both wrists
Central pain processing: dysfunctional endogenous pain analgesia | 1 year postoperative
  Measured with quantitative sensory testing (QST): conditioned pain modulation measured Medoc at both wrists
Central pain processing: somatic and emotional symptoms | Change from baseline (preoperative) to 3 months postoperative
  Questionnaire: the Central sensitization Inventory (CSI). Minimum score is 0, maximum score is 100. The higher the score, the higher the chance for the presence of central sensitization.
Central pain processing: somatic and emotional symptoms | Change from baseline (preoperative) to 1 year postoperative
  Questionnaire: the Central sensitization Inventory (CSI). Minimum score is 0, maximum score is 100. The higher the score, the higher the chance for the presence of central sensitization.
Central pain processing: somatic and emotional symptoms | Change from 3 months postoperative to 1 year postoperative
  Questionnaire: the Central sensitization Inventory (CSI). Minimum score is 0, maximum score is 100. The higher the score, the higher the chance for the presence of central sensitization.
Central pain processing: somatic and emotional symptoms | Baseline (preoperative)
  Questionnaire: the Central sensitization Inventory (CSI). Minimum score is 0, maximum score is 100. The higher the score, the higher the chance for the presence of central sensitization.
Central pain processing: somatic and emotional symptoms | 3 months postoperative
  Questionnaire: the Central sensitization Inventory (CSI). Minimum score is 0, maximum score is 100. The higher the score, the higher the chance for the presence of central sensitization.
Central pain processing: somatic and emotional symptoms | 1 year postoperative
  Questionnaire: the Central sensitization Inventory (CSI). Minimum score is 0, maximum score is 100. The higher the score, the higher the chance for the presence of central sensitization.
Central pain processing: areas of pain | Change from baseline (preoperative) to 3 months postoperative
  Body chart: Expanded distribution of Pain (EDP). The more pain locations, the more chance for the presence of central sensitization
Central pain processing: areas of pain | Change from baseline (preoperative) to 1 year postoperative
  Body chart: Expanded distribution of Pain (EDP). The more pain locations, the more chance for the presence of central sensitization
Central pain processing: areas of pain | Change from 3 months postoperative to 1 year postoperative
  Body chart: Expanded distribution of Pain (EDP). The more pain locations, the more chance for the presence of central sensitization
Central pain processing: areas of pain | Baseline (preoperative)
  Body chart: Expanded distribution of Pain (EDP). The more pain locations, the more chance for the presence of central sensitization
Central pain processing: areas of pain | 3 months postoperative
  Body chart: Expanded distribution of Pain (EDP). The more pain locations, the more chance for the presence of central sensitization
Central pain processing: areas of pain | 1 year postoperative
  Body chart: Expanded distribution of Pain (EDP). The more pain locations, the more chance for the presence of central sensitization
Psychosocial factors: pain catastrophizing | Change from baseline (preoperative) to 3 months postoperative
  Measured with Pain Catastrophizing Scale (PCS). Minimum score is 0, maximum score is 52. The higher the score, the higher the pain catastrophizing.
Psychosocial factors: pain catastrophizing | Change from baseline (preoperative) to 1 year postoperative
  Measured with Pain Catastrophizing Scale (PCS). Minimum score is 0, maximum score is 52. The higher the score, the higher the pain catastrophizing.
Psychosocial factors: pain catastrophizing | Change from 3 months postoperative to 1 year postoperative
  Measured with Pain Catastrophizing Scale (PCS). Minimum score is 0, maximum score is 52. The higher the score, the higher the pain catastrophizing.
Psychosocial factors: pain catastrophizing | Baseline (preoperative)
  Measured with Pain Catastrophizing Scale (PCS). Minimum score is 0, maximum score is 52. The higher the score, the higher the pain catastrophizing.
Psychosocial factors: pain catastrophizing | 3 months postoperative
  Measured with Pain Catastrophizing Scale (PCS). Minimum score is 0, maximum score is 52. The higher the score, the higher the pain catastrophizing.
Psychosocial factors: pain catastrophizing | 1 year postoperative
  Measured with Pain Catastrophizing Scale (PCS). Minimum score is 0, maximum score is 52. The higher the score, the higher the pain catastrophizing.
Psychosocial factors: illness perceptions | Change from baseline (preoperative) to 3 months postoperative
  Illness perception questionnaire-revised (IPQ-R)
  1. Identity dimension:
     yes = 1; no = 0 min score= 0, max score= 18
  2. Other dimensions:
     min score= 38, max score= 190 strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  3. Causal dimension:
  strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5 min score= 18, max score= 90
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.
Psychosocial factors: illness perceptions | Change from baseline (preoperative) to 1 year postoperative
  Illness perception questionnaire-revised (IPQ-R)
  1. Identity dimension:
     yes = 1; no = 0 min score= 0, max score= 18
  2. Other dimensions:
     min score= 38, max score= 190 strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  3. Causal dimension:
  strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5 min score= 18, max score= 90
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.
Psychosocial factors: illness perceptions | Change from 3 months postoperative to 1 year postoperative
  Illness perception questionnaire-revised (IPQ-R)
  1. Identity dimension:
     yes = 1; no = 0 min score= 0, max score= 18
  2. Other dimensions:
     min score= 38, max score= 190 strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  3. Causal dimension:
  strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5 min score= 18, max score= 90
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.
Psychosocial factors: illness perceptions | Baseline (preoperative)
  Illness perception questionnaire-revised (IPQ-R)
  1. Identity dimension:
     yes = 1; no = 0 min score= 0, max score= 18
  2. Other dimensions:
     min score= 38, max score= 190 strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  3. Causal dimension:
  strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5 min score= 18, max score= 90
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.
Psychosocial factors: illness perceptions | 3 months postoperative
  Illness perception questionnaire-revised (IPQ-R)
  1. Identity dimension:
     yes = 1; no = 0 min score= 0, max score= 18
  2. Other dimensions:
     min score= 38, max score= 190 strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  3. Causal dimension:
  strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5 min score= 18, max score= 90
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.
Psychosocial factors: illness perceptions | 1 year postoperative
  Illness perception questionnaire-revised (IPQ-R)
  1. Identity dimension:
     yes = 1; no = 0 min score= 0, max score= 18
  2. Other dimensions:
     min score= 38, max score= 190 strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5
  3. Causal dimension:
  strongly disagree =1, disagree =2, neither agree or disagree = 3, agree = 4, strongly agree = 5 min score= 18, max score= 90
  High scores on the identity, timeline, consequences, and cyclical dimensions represent strongly held beliefs about the number of symptoms attributed to the illness, the chronicity of the condition, the negative consequences of the illness, and the cyclical nature of the condition.
  High scores on the personal control, treatment control and coherence dimensions, represent positive beliefs about the controllability of the illness and a personal understanding of the condition.
Psychosocial factors: anxiety | Change from baseline (preoperative) to 3 months postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale anxiety. Minimum score is 0, maximum score is 21. The higher the score, the higher the anxiety.
Psychosocial factors: anxiety | Change from baseline (preoperative) to 1 year postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale anxiety. Minimum score is 0, maximum score is 21. The higher the score, the higher the anxiety.
Psychosocial factors: anxiety | Change from 3 months postoperative to 1 year postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale anxiety. Minimum score is 0, maximum score is 21. The higher the score, the higher the anxiety.
Psychosocial factors: anxiety | Baseline (preoperative)
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale anxiety. Minimum score is 0, maximum score is 21. The higher the score, the higher the anxiety.
Psychosocial factors: anxiety | 3 months postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale anxiety. Minimum score is 0, maximum score is 21. The higher the score, the higher the anxiety.
Psychosocial factors: anxiety | 1 year postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale anxiety. Minimum score is 0, maximum score is 21. The higher the score, the higher the anxiety.
Psychosocial factors: depression | Change from baseline (preoperative) to 3 months postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale depression. Minimum score is 0, maximum score is 21. The higher the score, the higher the depression.
Psychosocial factors: depression | Change from baseline (preoperative) to 1 year postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale depression. Minimum score is 0, maximum score is 21. The higher the score, the higher the depression.
Psychosocial factors: depression | Change from 3 months postoperative to 1 year postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale depression. Minimum score is 0, maximum score is 21. The higher the score, the higher the depression.
Psychosocial factors: depression | Baseline (preoperative)
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale depression. Minimum score is 0, maximum score is 21. The higher the score, the higher the depression.
Psychosocial factors: depression | 3 months postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale depression. Minimum score is 0, maximum score is 21. The higher the score, the higher the depression.
Psychosocial factors: depression | 1 year postoperative
  Measured with Hospital Anxiety and Depression Scale (HADS), subscale depression. Minimum score is 0, maximum score is 21. The higher the score, the higher the depression.
Functional factors: Maximal voluntary muscle strength m. Hamstrings | Change from baseline (preoperative) to 3 months postoperative
  Strength m. Hamstrings of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Hamstrings | Change from baseline (preoperative) to 1 year postoperative
  Strength m. Hamstrings of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Hamstrings | Change from 3 months postoperative to 1 year postoperative
  Strength m. Hamstrings of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Hamstrings | 3 months postoperative
  Strength m. Hamstrings of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Hamstrings | Baseline (preoperative)
  Strength m. Hamstrings of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Hamstrings | 1 year postoperative
  Strength m. Hamstrings of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Quadriceps | Change from baseline (preoperative) to 3 months postoperative
  Strength m. Quadriceps of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Quadriceps | Change from baseline (preoperative) to 1 year postoperative
  Strength m. Quadriceps of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Quadriceps | Change from 3 months postoperative to 1 year postoperative
  Strength m. Quadriceps of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Quadriceps | Baseline (preoperative)
  Strength m. Quadriceps of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Quadriceps | 3 months postoperative
  Strength m. Quadriceps of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: Maximal voluntary muscle strength m. Quadriceps | 1 year postoperative
  Strength m. Quadriceps of both legs, measured with Biodex System 4 pro - dynamometer
Functional factors: proprioceptive accuracy | Change from baseline (preoperative) to 3 months postoperative
  Proprioception of the knee of both legs, measured with inclinometer
Functional factors: proprioceptive accuracy | Change from baseline (preoperative) to 1 year postoperative
  Proprioception of the knee of both legs, measured with inclinometer
Functional factors: proprioceptive accuracy | Change from 3 months postoperative to 1 year postoperative
  Proprioception of the knee of both legs, measured with inclinometer
Functional factors: proprioceptive accuracy | Baseline (preoperative)
  Proprioception of the knee of both legs, measured with inclinometer
Functional factors: proprioceptive accuracy | 3 months postoperative
  Proprioception of the knee of both legs, measured with inclinometer
Functional factors: proprioceptive accuracy | 1 year postoperative
  Proprioception of the knee of both legs, measured with inclinometer
Functional factors: leg strength and endurance | Change from baseline (preoperative) to 3 months postoperative
  Measured with 30 seconds Timed Chair-Stand-Test
Functional factors: leg strength and endurance | Change from baseline (preoperative) to 1 year postoperative
  Measured with 30 seconds Timed Chair-Stand-Test
Functional factors: leg strength and endurance | Change from 3 months postoperative to 1 year postoperative
  Measured with 30 seconds Timed Chair-Stand-Test
Functional factors: leg strength and endurance | Baseline (preoperative)
  Measured with 30 seconds Timed Chair-Stand-Test
Functional factors: leg strength and endurance | 3 months postoperative
  Measured with 30 seconds Timed Chair-Stand-Test
Functional factors: leg strength and endurance | 1 year postoperative
  Measured with 30 seconds Timed Chair-Stand-Test
Patient demographics | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale patient demographics (nominal)
Alignment | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale objective knee score 'alignment': weight-bearing anterior-posterior radiograph measuring the femoral-tibial (Anatomic) axis. Minimum is 0, maximum is 25. The higher the score, the better the alignment.
Instability | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale objective knee score 'instability'. Minimum is 0, maximum is 25. The higher the score, the better the stability.
Joint motion | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale objective knee score 'joint motion'. Minimum is 0, maximum can be higher than 25. One point for every joint motion of 5 degrees. The higher the score, the better the joint motion.
Pain symptoms | Change from baseline (preoperative) to 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale symptoms. Minimum score is 0, maximum score is 25. The higher the score, the worse the pain symptoms.
Pain symptoms | Change from baseline (preoperative) to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale symptoms. Minimum score is 0, maximum score is 25. The higher the score, the worse the pain symptoms.
Pain symptoms | Change from 3 months postoperative to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale symptoms. Minimum score is 0, maximum score is 25. The higher the score, the worse the pain symptoms.
Pain symptoms | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale symptoms. Minimum score is 0, maximum score is 25. The higher the score, the worse the pain symptoms.
Pain symptoms | 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale symptoms. Minimum score is 0, maximum score is 25. The higher the score, the worse the pain symptoms.
Pain symptoms | 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale symptoms. Minimum score is 0, maximum score is 25. The higher the score, the worse the pain symptoms.
Patient expectations | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale patient expectations. Minimum score is 0, maximum score is 15. The higher the score, the higher the patient's opinion on the extent to which the patient expects that the operation will improve their knee pain, and their ability to perform their activities of daily living and recreational activities
Patient expectations fulfillment | 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale patient expectations. Minimum score is 0, maximum score is 15. The higher the score, the higher the patient's opinion on the extent to which the outcome after the operation has met the patient's pre-operative expectations with respect to pain and function
Patient expectations fulfillment | 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale patient expectations. Minimum score is 0, maximum score is 15. The higher the score, the higher the patient's opinion on the extent to which the outcome after the operation has met the patient's pre-operative expectations with respect to pain and function
Patient expectations fulfillment | Change from 3 months postoperative to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale patient expectations. Minimum score is 0, maximum score is 15. The higher the score, the higher the patient's opinion on the extent to which the outcome after the operation has met the patient's pre-operative expectations with respect to pain and function
Patient satisfaction | Change from baseline (preoperative) to 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale patient satisfaction. Minimum score is 0, maximum score is 40. The higher the score, the more satisfied the patient feels with their knee.
Patient satisfaction | Change from baseline (preoperative) to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale patient satisfaction. Minimum score is 0, maximum score is 40. The higher the score, the more satisfied the patient feels with their knee.
Patient satisfaction | Change from 3 months postoperative to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale patient satisfaction. Minimum score is 0, maximum score is 40. The higher the score, the more satisfied the patient feels with their knee.
Patient satisfaction | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale patient satisfaction. Minimum score is 0, maximum score is 40. The higher the score, the more satisfied the patient feels with their knee.
Patient satisfaction | 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale patient satisfaction. Minimum score is 0, maximum score is 40. The higher the score, the more satisfied the patient feels with their knee.
Patient satisfaction | 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale patient satisfaction. Minimum score is 0, maximum score is 40. The higher the score, the more satisfied the patient feels with their knee.
Functional score | Change from baseline (preoperative) to 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale functional score. Minimum score is 0, maximum score is 100. The higher the score, the better the functionality of the patient
Functional score | Change from baseline (preoperative) to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale functional score. Minimum score is 0, maximum score is 100. The higher the score, the better the functionality of the patient
Functional score | Change from 3 months postoperative to 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale functional score. Minimum score is 0, maximum score is 100. The higher the score, the better the functionality of the patient
Functional score | Baseline (preoperative)
  measured with Knee Society Scoring System (KSS): subscale functional score. Minimum score is 0, maximum score is 100. The higher the score, the better the functionality of the patient
Functional score | 3 months postoperative
  measured with Knee Society Scoring System (KSS): subscale functional score. Minimum score is 0, maximum score is 100. The higher the score, the better the functionality of the patient
Functional score | 1 year postoperative
  measured with Knee Society Scoring System (KSS): subscale functional score. Minimum score is 0, maximum score is 100. The higher the score, the better the functionality of the patient
Metabolic factors: Fat mass | Change from baseline (preoperative) to 3 months postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Fat mass | Change from baseline (preoperative) to 1 year postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Fat mass | Change from 3 months postoperative to 1 year postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Fat mass | Baseline (preoperative)
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Fat mass | 3 months postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Fat mass | 1 year postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Lean mass | Change from baseline (preoperative) to 3 months postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Lean mass | Change from baseline (preoperative) to 1 year postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Lean mass | Change from 3 months postoperative to 1 year postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Lean mass | Baseline (preoperative)
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Lean mass | 3 months postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Lean mass | 1 year postoperative
  Measured with Bio-electrical Impedance Analyses (BIA)
Metabolic factors: Body mass index (BMI) | Change from baseline (preoperative) to 3 months postoperative
  Measured with length of patient (cm) and weight of patient (kg)
Metabolic factors: Body mass index (BMI) | Change from baseline (preoperative) to 1 year postoperative
  Measured with length of patient (cm) and weight of patient (kg)
Metabolic factors: Body mass index (BMI) | Change from 3 months postoperative to 1 year postoperative
  Measured with length of patient (cm) and weight of patient (kg)
Metabolic factors: Body mass index (BMI) | Baseline (preoperative)
  Measured with length of patient (cm) and weight of patient (kg)
Metabolic factors: Body mass index (BMI) | 3 months postoperative
  Measured with length of patient (cm) and weight of patient (kg)
Metabolic factors: Body mass index (BMI) | 1 year postoperative
  Measured with length of patient (cm) and weight of patient (kg)
Metabolic factors: body composition | Baseline (preoperative), 3 months postoperative, 1 year postoperative.
  Measured with Bioelectrical Impedance Analysis (BIA)
Metabolic factors: venous blood sample | Change from baseline (preoperative) to 3 months postoperative
  Measured with A1C test or glycohemoglobin test
Metabolic factors: venous blood sample | Change from baseline (preoperative) to 1 year postoperative
  Measured with A1C test or glycohemoglobin test
Metabolic factors: venous blood sample | Change from 3 months postoperative to 1 year postoperative
  Measured with A1C test or glycohemoglobin test
Metabolic factors: venous blood sample | Baseline (preoperative)
  Measured with A1C test or glycohemoglobin test
Metabolic factors: venous blood sample | 3 months postoperative
  Measured with A1C test or glycohemoglobin test
Metabolic factors: venous blood sample | 1 year postoperative.
  Measured with A1C test or glycohemoglobin test
Structural factors | Baseline (preoperative)
  Measured with Kellgren and Lawrence scale on radiography
Inflammatory factors: signs of inflammation | Baseline (preoperative)
  Measured with the C-reactive protein levels in blood sample (collected from patient record)
Anesthetic procedure | During surgery
  General anesthesia, spinal anesthesia or combination with peripheral block
Clinical pain score | day 1 and 2 postoperative
  Measured with numeric rating pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Vervullens, Principal Investigator — Universiteit Antwerpen; Lotte Meert, Principal Investigator — Universiteit Antwerpen; Mira Meeus, Principal Investigator — Universiteit Antwerpen; Isabel Baert, Principal Investigator — Universiteit Antwerpen; Rob J.E.M. Smeets, Principal Investigator — Maastricht University
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vervullens S, Meert L, Smeets RJEM, van der Nest G, Verbrugghe J, Verdonk P, Rahusen FTG, Meeus M. A biopsychosocial approach to phenotyping people with knee osteoarthritis awaiting total knee arthroplasty: A secondary cohort analysis. Ann Phys Rehabil Med. 2024 Nov;67(8):101895. doi: 10.1016/j.rehab.2024.101895. Epub 2024 Oct 28. PMID 39489935
- [Derived] Vervullens S, Meert L, Smeets RJEM, Verbrugghe J, Baert I, Rahusen FTG, Heusdens CHW, Verdonk P, Meeus M. Preoperative glycaemic control, number of pain locations, structural knee damage, self-reported central sensitisation, satisfaction and personal control are predictive of 1-year postoperative pain, and change in pain from pre- to 1-year posttotal knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2025 Jan;33(1):201-219. doi: 10.1002/ksa.12265. Epub 2024 May 15. PMID 38751081
- [Derived] Vervullens S, Meert L, Smeets RJEM, Verbrugghe J, Verdonk P, Meeus M. Does pain intensity after total knee arthroplasty depend on somatosensory functioning in knee osteoarthritis patients? A prospective cohort study. Clin Rheumatol. 2024 Jun;43(6):2047-2059. doi: 10.1007/s10067-024-06976-7. Epub 2024 Apr 26. PMID 38668988